CLINICAL TRIAL: NCT05585788
Title: Efficacy of a Pill-Dispensing System to Increase Disposal of Unused Opioids and to Reduce Refills After Cancer-Related Surgery
Brief Title: Opioid Dispensing Device for Post-Operative Pain in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Assistant Professor of Medicine, Division of Hematology/Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAS8214
Record Dates: First submitted 2022-03-09; First posted 2022-10-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: To assess the impact of a password-protected pill-dispensing system, Addinex, on unused opioid disposal, opioid use, and opioid refills rates after cancer-related surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Addinex system (Other): The Addinex system is designed to dispense opioid medication to patients on a provider-determined schedule, to track patient use of the device, and to allow for return and disposal of unused opioids. This study will determine the feasibility of using Addinex for these purposes.
  Interventions: Device: Addinex Device (ADX-27)

INTERVENTIONS:
Device: Addinex Device (ADX-27) — The device operates without the use of any electronics, wireless or firmware requirements. This is achieved through its mechanical system which uses a different randomized "passcode" for each dose that is loaded into a circular drum inside the device. The "passcodes" are provided by an online server through either a mobile app, web app, text service or call in service. The online server provides "passcodes" on a request basis, while following instructions set by the treating physicians.

SUMMARY:
This research study will evaluate the use of, and participants experience with, a new device called Addinex that safely stores and dispenses opioid medication. The purpose of this study is to evaluate the use of the Addinex device in cancer patients undergoing cancer-related surgery that require pain control with opioids after the surgery. Participants will be asked to answer questions about their medical history and background, fill out questionnaires, use a mobile application associated with the device, and undergo a phone interview one month after stopping use of the device. This study aims to find out how participants like using the Addinex device as opposed to a traditional pill bottle. Results of this study will help determine if the Addinex device could be useful to patients in the future after surgeries, as opposed to typical pill bottles.

DETAILED DESCRIPTION:
This is a non-randomized pilot study to test the use of the Addinex system among participants receiving opioids following surgery. The Addinex system is designed to dispense opioid medication to participants on a provider-determined schedule, to track participant use of the device, and to allow for return and disposal of unused opioids. This study will determine the feasibility of using Addinex for these purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age greater than or equal to 18 years)
* Planned for major cancer-related surgery and expected to receive a postoperative opioid prescription
* Must speak English or Spanish
* Must have access to a smartphone or an alternative smart device (e.g., iPhone, Android phone, iPad, Surface, etc.).
* Co-enrollment in trials involving pharmacologic therapy is allowed

Exclusion Criteria:

* Patients who are taking opioids daily prior to the surgical procedure
* Patients unable to physically utilize the device
* Patients unable to self-administer medications
* Patients uncomfortable with using iPhone or iPad-based technology

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Device Return | 12 weeks
  The rate of device return will be determined by an online logging of returned devices by a medical waste disposal company.
Rate of Unused Pill Disposal | 12 weeks
  The number of unused pills disposed will be deduced based on the number of passwords requested from returned devices.

SECONDARY OUTCOMES:
Median Pill Consumption | 12 weeks
  Median opioid consumption will be deduced from the number of password requests. Number, date and time of participant password requests are logged on an online database maintained by Addinex.
Duration of Opioid Use | 12 weeks
  Opioid Use Duration will be measured in days and deduced from the dates of password requests. Number, date and time of participant password requests are logged on an online database maintained by Addinex.
Opioid Refill Rate | 12 weeks
  Opioid refill rates will be determined through review of electronic medical records and state prescription monitoring programs.
Change in Brief Pain Inventory (BPI) Score Baseline and 3 Days | Baseline and Day 3
  The quality of pain control will be measured using BPI, which measures two domains: pain severity and pain interference on daily activities. Scores range from 0 to 10 with lower score indicating a better outcome.
Change in Brief Pain Inventory (BPI) Score Baseline and 7 Days | Baseline and Day 7
  The quality of pain control will be measured using BPI, which measures two domains: pain severity and pain interference on daily activities. Scores range from 0 to 10 with lower score indicating a better outcome.
Change in Brief Pain Inventory (BPI) Score Baseline and 3 Weeks | Baseline and Week 3
  The quality of pain control will be measured using BPI, which measures two domains: pain severity and pain interference on daily activities. Scores range from 0 to 10 with lower score indicating a better outcome.
Post Study System Usability Questionnaire (PSSUQ) Score | 3 weeks
  Device usability will be measured by the PSSUQ questionnaire, a 19-item scale. Scores range from 1 (strongly agree) to 7 (strongly disagree) with lower score indicating greater usability.
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) Scores | 3 weeks
  Acceptability, appropriateness, and feasibility will be measured by combining AIM, IAM, and FIM scale scores. The combination of these scales demonstrates strong psychometric properties and is being used in other cancer-related and technology-based intervention research. Scores range from 1 (Strongly Disagree) to 5 (Completely Agree) with a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No